CLINICAL TRIAL: NCT02643979
Title: Ketamine and Propofol Combination Versus Propofol for Upper Gastrointestinal Endoscopy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GCO 15-2139
Record Dates: First submitted 2015-12-22; First posted 2015-12-31 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Bariatrics; Sleep Apnea Syndromes; Gastric Bypass; Endoscopy
Keywords: Ketamine; Propofol; Ketofol; Obese; Upper gastrointestinal endoscopy; Sedation; Bariatric
MeSH Terms: conditions — Obesity; Sleep Apnea Syndromes | interventions — Ketamine; Propofol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketofol and Propofol (Experimental): This arm receives a 50mg dose of Ketamine mixed with 100mg of Propofol at the start of their upper endoscopy.
  Interventions: Drug: Ketofol; Drug: Propofol
- Propofol only (Active Comparator): This arm receives 100mg of Propofol mixed with 1mL of saline at the start of the upper gastrointestinal endoscopy.
  Interventions: Drug: Propofol; Drug: Saline

INTERVENTIONS:
Drug: Ketofol — 50mg of Ketamine mixed with 100mg of Propofol
  Other Names: Ketamine and Propofol; Ketalar; Diprivan
  Arms: Ketofol and Propofol
Drug: Propofol — 100mg of Propofol
  Other Names: Diprivan
Drug: Saline — 1mL of saline
  Arms: Propofol only

SUMMARY:
Propofol is one of the most popular anesthetic drugs used for sedation during upper gastrointestinal endoscopies due to its quick onset and quick resolution of symptoms allowing patients to leave the hospital sooner. However, when administered it can also slow the breathing of patients and cause others to have upper airway obstruction (such as snoring) which can impede proper spontaneous breathing. Ketamine is an agent that is capable of providing both pain control and sedation while having either minimal effect on breathing or promoting spontaneous breathing. Combining Ketamine with Propofol has the potential to reduce the total amount of Propofol used resulting in a procedure being performed under the same level of sedation but without the downside of reduced spontaneous breathing. Patients who are obese (defined as body mass index greater than 35) tend to be even more susceptible to this effect of Propofol. The researchers are investigating whether the addition of Ketamine will indeed allow for this continued comfortable level of sedation while promoting continued spontaneous breathing in obese patients undergoing upper gastrointestinal endoscopies.

DETAILED DESCRIPTION:
Upon patient arrival to endoscopy suite heart rate (HR), pre-procedure baseline blood pressure (BP), and pre-procedure oxygen saturation (SPO2) via pulse oximeter are recorded in endoscopy holding area, patient alertness and orientation assessed (respond to name, know the state, know the hospital, know the year, know the season).

Once the subject enters the endoscopy suite monitors are placed to record starting BP, HR, SPO2 recorded, nasal cannula with end tidal carbon dioxide (CO2) monitor attached, and 5-lead ECG.

Following time out patient given 100mg Lidocaine IV bolus, 1-minute delay, then study-provided syringe administered. Once patient assessed to produce an RSS score >5 (Asleep with sluggish response to glabellar tap or NO response) endoscopy proceeds.

Recorder (blinded) notes if initially provided syringe alone was enough to produce an RSS >5, notes subject's response to endoscopy insertion (presence or absence of gagging), notes amount of additional propofol required to maintain adequate conditions to continue endoscopy, records non-invasive blood pressure (NIBP) at 3-minute intervals, notes for level of airway obstruction (obstruction with continued air movement, obstruction requiring chin lift or jaw thrust for relief, obstruction requiring progression to assisted ventilation or intubation), notes for desaturation events (SPO2 <90% with a coherent waveform).

At the end of the procedure the total anesthesia time is recorded, total procedure start-to-finish time recorded, total dose of propofol recorded, and any incidence of patient agitation noted.

Once in recovery the recovery room admission HR, SPO2, NIBP recorded followed by admission +15 minutes HR, SPO2, and NIBP, any incidence of desaturation (<90% SPO2 with waveform) recorded, incidence of airway obstruction (with air movement, requiring airway maneuver, requiring intervention) recorded, time until patient is alert and oriented recorded (response to name, able to state what state they are in, able to state what hospital they are in, able to state the year, able to state the season), time-until-recovered recorded (Modified Aldrete Score > 9), incidence of nausea prior to recovery recorded, incidence of vomiting prior to recovery recorded, incidence of agitation or delirium prior to recovery recorded.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30
* Undergoing an upper gastrointestinal endoscopy

Exclusion Criteria:

* History of schizophrenia/schizoaffective disorder
* History of bipolar disorder
* History of dementia
* Non-English Speaking
* History of Glaucoma
* Craniofacial Abnormalities
* Epilepsy
* Allergy to Propofol
* Allergy to Ketamine
* Current known intracranial mass/lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Katz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; David A Maerz, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tandon M, Pandey VK, Dubey GK, Pandey CK, Wadhwa N. Addition of sub-anaesthetic dose of ketamine reduces gag reflex during propofol based sedation for upper gastrointestinal endoscopy: A prospective randomised double-blind study. Indian J Anaesth. 2014 Jul;58(4):436-41. doi: 10.4103/0019-5049.138981. PMID 25197112
- [Background] Dal T, Sazak H, Tunc M, Sahin S, Yilmaz A. A comparison of ketamine-midazolam and ketamine-propofol combinations used for sedation in the endobronchial ultrasound-guided transbronchial needle aspiration: a prospective, single-blind, randomized study. J Thorac Dis. 2014 Jun;6(6):742-51. doi: 10.3978/j.issn.2072-1439.2014.04.10. PMID 24976998
- [Background] Street MH, Gerard JM. A fixed-dose ketamine protocol for adolescent sedations in a pediatric emergency department. J Pediatr. 2014 Sep;165(3):453-8. doi: 10.1016/j.jpeds.2014.03.021. Epub 2014 Apr 20. PMID 24755240
- [Background] Newton A, Fitton L. Intravenous ketamine for adult procedural sedation in the emergency department: a prospective cohort study. Emerg Med J. 2008 Aug;25(8):498-501. doi: 10.1136/emj.2007.053421. PMID 18660398
- [Background] Sih K, Campbell SG, Tallon JM, Magee K, Zed PJ. Ketamine in adult emergency medicine: controversies and recent advances. Ann Pharmacother. 2011 Dec;45(12):1525-34. doi: 10.1345/aph.1Q370. Epub 2011 Dec 6. PMID 22147144
- [Background] Pambianco DJ. Future directions in endoscopic sedation. Gastrointest Endosc Clin N Am. 2008 Oct;18(4):789-99, x. doi: 10.1016/j.giec.2008.06.004. PMID 18922416

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketofol: Ketamine and Propofol: This arm received a 50mg dose of Ketamine mixed with 100mg of Propofol at the start of their upper endoscopy.
- Propofol Only: This arm received 100mg of Propofol mixed with 1mL of saline at the start of the upper gastrointestinal endoscopy.
Period: Overall Study
Arm/Group | Ketofol: Ketamine and Propofol | Propofol Only
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketofol: Ketamine and Propofol | Propofol Only | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.09 (16.0) | 44.63 (9.39) | 48.86 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 41 (5.4) | 44 (8.3) | 42.5 (7.2)
ASA Class [Mean (Standard Deviation); unit: units on a scale] — American Society of Anesthesiologists Classification (ASA Class)
  ASA 1 A normal healthy patient
  ASA 2 A patient with mild systemic disease
  ASA 3 A patient with severe systemic disease
  ASA 4 A patient with severe systemic disease that is a constant threat to life
  ASA 5 A moribund patient who is not expected to survive without the operation
  ASA 6 A declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 2.9 (0.2) | 3 (0) | 2.9 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Gagging Reaction
Description: Number of participants with gagging or "vomit-like" reaction on endoscopic insertion
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ketofol: Ketamine and Propofol | Propofol Only
Number analyzed (Participants) | 11 | 11
Participants | 2 | 1

2. Secondary Outcome: Number of Participants With Any Type of Airway Obstruction
Description: The Anesthesiologist caring for the patient during the upper endoscopy made note of any obstructive events defined on a scale ranging from the patient audibly snoring (obstructing) to the patient obstructing and requiring assistance such as a chin lift or jaw thrust to relieve the obstruction and continue to move air adequately.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ketofol: Ketamine and Propofol | Propofol Only
Number analyzed (Participants) | 11 | 11
Participants | 4 | 3

3. Secondary Outcome: Total Dose of Propofol Used During the Procedure
Description: Propofol doses are logged in the computerized Compurecord system used in the operating room. Patients involved in the study had their total Propofol dose required quantified and compared between groups who received Ketamine and groups who did not.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Ketofol: Ketamine and Propofol | Propofol Only
Number analyzed (Participants) | 11 | 11
mg/kg | 9.09 (19) | 39 (57.3)

4. Secondary Outcome: Total Sedation Required to Allow Initiation of Procedure
Description: Using the computerized record system, the amount of Propofol a patient required to allow for the procedure to start quantified and compared between groups.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Ketofol: Ketamine and Propofol | Propofol Only
Number analyzed (Participants) | 11 | 11
mg/kg | 78 (50.6) | 61 (57.2)

5. Secondary Outcome: Number of Participants With Post-operative Nausea and/or Vomiting
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ketofol: Ketamine and Propofol | Propofol Only
Number analyzed (Participants) | 11 | 11
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Emergence Delirium
Description: Number of participants with emergence delirium measured from the procedure end until time of discharge.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ketofol: Ketamine and Propofol | Propofol Only
Number analyzed (Participants) | 11 | 11
Participants | 0 | 0

7. Secondary Outcome: Time to Recovery
Description: Monitored via the electronic medical record system as the time between the anesthesia end time and when the patient was safe for discharge from the hospital.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ketofol: Ketamine and Propofol | Propofol Only
Number analyzed (Participants) | 11 | 11
minutes | 21 (9) | 25 (5)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Ketofol and Propofol: This arm received a 50mg dose of Ketamine mixed with 100mg of Propofol at the start of their upper endoscopy.
Arm/Group | Ketofol and Propofol | Propofol Only
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-08-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT02643979/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT02643979/SAP_001.pdf